CLINICAL TRIAL: NCT04744818
Title: Effects of Iron Supplementation on Pediatric Vaccine Response
Acronym: VINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessica Rigutto (Other)
Collaborators: Jomo Kenyatta University of Agriculture and Technology Kenya (Unknown); Karolinka Institute Sweden (Unknown); University of Oxford (Other); National Institute for Public Health and Environment Netherlands (Unknown)
Responsible Party: Sponsor-Investigator, Jessica Rigutto, Dr. Nicole Stoffel, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: VINO
Record Dates: First submitted 2021-01-28; First posted 2021-02-09 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia; Vaccination; Pediatric ALL
MeSH Terms: conditions — Anemia, Iron-Deficiency; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate iron treatment (Active Comparator): Iron and multivitamin syrup
  Interventions: Dietary Supplement: Iron syrup; Dietary Supplement: Multivitamin syrup
- Delayed iron treatment (Placebo Comparator): Multivitamin syrup
  Interventions: Dietary Supplement: Multivitamin syrup

INTERVENTIONS:
Dietary Supplement: Iron syrup — Daily supplementation with iron
  Arms: Immediate iron treatment
Dietary Supplement: Multivitamin syrup — Daily supplementation with multivitamins

SUMMARY:
ID/IDA affects many young children in Africa. Vaccines provide tremendous benefits in LMIC; however, they currently fail to reach their full potential. We need to better understand the causes of vaccine failure, in order to develop new strategies to improve vaccine immunogenicity.

This study will contribute to children's health by: (1) providing updated guidelines to better define the prevalence of ID/IDA in early infancy, and its safe and effective control using iron; and (2) providing a new approach to improve response to pediatric vaccines in LMIC, by ensuring adequate iron status at time of vaccination.

DETAILED DESCRIPTION:
Two major pediatric public health goals in LMIC are increasing immunization effectiveness and reducing ID/IDA in children. ID/IDA affects many young children in Africa. Current guidelines do not recommend routine testing of hemoglobin in early infancy, as it is generally believed that most infants are born with adequate iron stores to last 6 months. However, many African infants are born with low iron stores and ID/IDA may develop earlier than generally appreciated, within 2-3 months after birth. Vaccines provide tremendous benefits in LMIC; however, they currently fail to reach their full potential. We need to better understand the causes of vaccine failure, in order to develop new strategies to improve vaccine immunogenicity. Despite lower efficacy in LMIC, these vaccines provide a major benefit because the disease burden is so high; however, if approaches can be found to improve immunogenicity, these vaccines would be even more powerful.

For this study, 6 weeks old infants will be randomly assigned to two study groups. Group 1 will receive iron at time of pediatric vaccinations from age 6-24 weeks. Group 2 will receive no iron at time of pediatric vaccinations. All infants will receive a multivitamin syrup from age 6-24 weeks. All infants remaining ID/IDA at age 24 weeks will receive iron. Infants will be followed-up until age 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Mother at least ≥15 years of age.
* 6 weeks (+/- 3 days) of age
* Iron deficient (erythrocyte zinc protoporphyrin (ZnPP) >61 μmol/mol heme)
* With or without anemia, but not severely anemic (Hb >70 g/L)
* No malaria
* No medical condition that precludes study involvement
* Mother HIV negative
* Vaginal delivery
* No iron supplementation prior to study enrolment
* Not wasted (length for height z score of ≥-2)
* Not underweight (weight for age z score ≥-2)
* From the hospital record, term or late preterm delivery (≥34 weeks)
* Full-time breastfed at least until the screening
* No vaccines beyond the birth dose of OPV and BCG prior to enrolment

Ages: 39 Days to 45 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 288 (Actual)
Dates: Start 2021-02-07 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Pertussis antibody profile | from 6 to 24 weeks
Diphtheria antibody profile | from 6 to 24 weeks

SECONDARY OUTCOMES:
antiviral immunoglobulin G response | 6 weeks of age
  Immunoassay
antiviral immunoglobulin G response | 24 weeks of age
  Immunoassay
infant antiviral immunoglobulin G response | 52 weeks of age
  Immunoassay
immune cell populations | 6 weeks of age
  number and type of immune cells
immune cell populations | 24 weeks of age
  number and type of immune cells
immune cell populations | 52 weeks of age
  number and type of immune cells
Proteomics | 6 weeks of age
  Proteins involved in immune response
Proteomics | 24 weeks of age
  Proteins involved in immune response
Proteomics | 52 weeks of age
  Proteins involved in immune response
Transcriptomics | 24 weeks of age
  Genes involved in immune response
Intestinal fatty acid binding protein | 6 weeks of age
  Gut inflammation
Intestinal fatty acid binding protein | 14 weeks of age
  Gut inflammation
Intestinal fatty acid binding protein | 24 weeks of age
  Gut inflammation
Calprotectin | 6 weeks of age
  Gut inflammation
Calprotectin | 14 weeks of age
  Gut inflammation
Calprotectin | 24 weeks of age
  Gut inflammation
Hemoglobin | 6 weeks of age
Hemoglobin | 14 weeks of age
Hemoglobin | 24 weeks of age
Hemoglobin | 38 weeks of age
Hemoglobin | 52 weeks of age
Plasma iron | 6 weeks of age
Plasma iron | 14 weeks of age
Plasma iron | 24 weeks of age
Plasma iron | 38 weeks of age
Plasma iron | 52 weeks of age
Plasma ferritin | 6 weeks of age
Plasma ferritin | 14 weeks of age
Plasma ferritin | 24 weeks of age
Plasma ferritin | 38 weeks of age
Plasma ferritin | 52 weeks of age
soluble transferrin receptor | 6 weeks of age
soluble transferrin receptor | 14 weeks of age
soluble transferrin receptor | 24 weeks of age
soluble transferrin receptor | 38 weeks of age
soluble transferrin receptor | 52 weeks of age
C-reactive protein | 6 weeks of age
C-reactive protein | 14 weeks of age
C-reactive protein | 24 weeks of age
C-reactive protein | 38 weeks of age
C-reactive protein | 52 weeks of age
Alpha-glycoprotein | 6 weeks of age
Alpha-glycoprotein | 14 weeks of age
Alpha-glycoprotein | 24 weeks of age
Alpha-glycoprotein | 38 weeks of age
Alpha-glycoprotein | 52 weeks of age
Tetanus antibody profile | from 6 to 24 weeks
Haemophilus influenzae b antibody profile | from 6 to 24 weeks
Pneumococcus antibody profile | from 6 to 24 weeks
Rotavirus antibody profile | from 6 to 24 weeks
Polio antibody profile | from 6 to 24 weeks
Anti-vaccine antibody titers | 38 weeks of age
Anti-vaccine antibody titers | 52 weeks of age
Anti-vaccine seroconversion | 14 weeks of age
Anti-vaccine seroconversion | 24 weeks of age
Anti-vaccine seroconversion | 38 weeks of age
Anti-vaccine seroconversion | 52 weeks of age
Anti-vaccine antibody avidity index | 14 weeks of age
  percentage of antibodies that remain bound to beads
Anti-vaccine antibody avidity index | 24 weeks of age
  percentage of antibodies that remain bound to beads
Anti-vaccine antibody avidity index | 38 weeks of age
  percentage of antibodies that remain bound to beads
Anti-vaccine antibody avidity index | 52 weeks of age
  percentage of antibodies that remain bound to beads

OTHER OUTCOMES:
Human milk oligosaccharide secretor type | 14 weeks of age
  secretor yes or no
Erythrocyte zinc protoporphyrin | 6 weeks of age
Erythrocyte zinc protoporphyrin | 14 weeks of age
Erythrocyte zinc protoporphyrin | 24 weeks of age
Erythrocyte zinc protoporphyrin | 38 weeks of age
Erythrocyte zinc protoporphyrin | 52 weeks of age

CONTACTS AND LOCATIONS:
Locations (2):
- Msambweni County Referral Hospital, Msambweni, Kwale County, Kenya
- Human Nutrition Laboratory ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No